CLINICAL TRIAL: NCT03360994
Title: Assessment of the WATChmAN (Web virtuAl Testicular CANcer Clinic): A Randomized Controlled Study to Estimate the Efficacy of an Electronic Surveillance Tool for Stage I Testicular Cancer
Brief Title: WATChmAN Virtual Testicular Cancer Clinic
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 17-5366
Record Dates: First submitted 2017-11-27; First posted 2017-12-04 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Testicular Cancer
MeSH Terms: conditions — Testicular Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WATChmAN (Experimental): Patients randomized to the WATChmAN Active Surveillance arm will receive their active surveillance testicular cancer care via an online virtual clinic. Importantly, patients will follow the same surveillance schedule as patients in the standard of care arm. However, patients in the WATChmAN arm will be able to see their upcoming tests and virtual appointments online, request requisitions to perform their required testing at outside institutions, and indicate any concerns for physicians to review during the virtual visit.
  Interventions: Other: WATChmAN Active Surveillance
- Standard of Care (Active Comparator): Patients randomized to the standard of care arm (in-person active surveillance) will follow the current active surveillance protocol in place at Princess Margaret Cancer Centre's Multidisciplinary Testicular Cancer Clinic. This protocol involves the same schedule of testing as the WATChmAN arm, but will require patients to come into the clinic to receive their test results (as in current practice).
  Interventions: Other: In-person Active Surveillance

INTERVENTIONS:
Other: WATChmAN Active Surveillance — WATChmAN Active Surveillance uses an electronic tool used to provide active surveillance care to testicular cancer patients. This virtual active surveillance care is delivered with an identical schedule to in-person care without the need to come into clinic.
  Arms: WATChmAN
Other: In-person Active Surveillance — In-person active surveillance is the current recommended management option for all Stage I testicular cancer patients at Princess Margaret. Patients are monitored clinically with imaging and blood work, and active treatment only begins if relapse occurs.
  Arms: Standard of Care

SUMMARY:
Princess Margaret's Multidisciplinary Testicular Cancer (TCa) Clinic sees over 25% of Ontario's testicular cancer patients, many of whom travel long distances. Fortunately, the majority of cases are confined to the testicle and are managed by "active surveillance" (AS), whereby blood work and imaging at regular intervals look to detect relapse at a curable stage. This currently requires multiple clinic visits over 5-9 years. This follow-up can be time-consuming, costly, difficult to adhere to and unsatisfying for patients. The goal of this project is to develop an efficient technological platform to perform virtual cancer follow-up. The platform has been named, "WATChmAN" which stands for Web-based virtual Testicular CANcer clinic. It will provide a secure, online interface to all virtual follow-up visits as an alternative to costly and time-consuming travel for in-person visits. The investigators anticipate improved patient satisfaction and dramatic reductions in the cost of cancer care follow-up. Moreover, the investigators anticipate improved compliance, which will lead to safer care. While TCa serves as the working platform, the investigators envision the end-product to be scalable and generalizable to other cancers (e.g. prostate cancer surveillance) across the province.

DETAILED DESCRIPTION:
Patients randomized to the standard of care arm will be required to follow the active surveillance protocol created by the Multidisciplinary Testicular Cancer Clinic at Princess Margaret Hospital. This involves blood marker and CT tests at predetermined intervals for 5-9 years depending on the patient's testicular cancer diagnosis (seminoma vs. non-seminoma). If randomized to this group, participants will be required to return to the Multidisciplinary Testicular Cancer Clinic to receive the results of their surveillance testing face-to-face in a medical appointment. In addition to these surveillance testing and follow-up visits, participants will also be asked to complete surveys regarding their satisfaction with the in-person active surveillance program. These surveys will take approximately 10-15 minutes to complete and will be predominantly multiple choice. These surveys will be emailed to participants at 6 months, 1 year, 2 years and 5 years after the study begins. As per current standard of care practice, participants may choose to have their imaging completed at a centre outside of the UHN. In these cases, participants will be required to obtain and send CDs with their imaging and reports to their most responsible oncologist at Princess Margaret. Blood marker visits can be performed anywhere without sending the results to Princess Margaret.

Patients randomized to the WATChmAN group will also be required to follow the active surveillance protocol created by the Multidisciplinary Testicular Cancer Clinic at Princess Margaret Hospital. If randomized to this group, a physician from the Multidisciplinary Testicular Cancer Clinic will still review the participant's surveillance testing results but will interact with the WATChmAN platform instead of receiving their results face-to-face in a medical appointment. Specifically, if randomized to this group participants will be required to:

* Asked, but not required, to have their picture taken to be uploaded into the WATChmAN platform. Their photo will only be stored on the password-protected WATChmAN database and will serve to cue facial recognition in the physicians reviewing their results and therefore enhance recall of their personal history.
* Confirm their registration in the WATChmAN program via a welcome email
* Respond to WATChmAN generated messages and reminders requesting whether or not their upcoming surveillance testing (e.g. blood tests and/or CT imaging scans) has been completed
* Respond to WATChmAN generated messages to confirm where their upcoming testing (e.g. blood tests and/or CT imaging scans) has been completed
* Check their results on the WATChmAN platform and express any concerns/issues they might have about their treatment and/or health to their most responsible oncologist through the WATChmAN platform
* Confirm receipt of messages concerning whether they need or do not need to come in for an in-person follow up visit
* Return to the Multidisciplinary Testicular Cancer Clinic to see a physician face-to-face for a final exit follow-up appointment when their active surveillance treatment is complete
* If getting their CT imaging visits outside the UHN, obtain and send CDs with their imaging and reports to the WATChmAN research coordinator for upload into the WATChmAN system (please note: this requirement is identical for patients in the standard of care group)
* Participants do not need to send in their blood test results. Their blood marker visits can be performed anywhere without needing to send them to the WATChmAN coordinator.

Finally, in addition to these surveillance testing and WATChmAN interactions, participants will also be asked to complete surveys regarding their satisfaction with their virtual active surveillance program. These surveys will take approximately 10-15 minutes to complete and will be predominantly multiple choice. These surveys will be emailed to participants at 6 months, 1 year, 2 years and 5 years after the study begins.

It is predicted that the WATChmAN virtual platform will take at least one year to construct; however, the researchers involved in this study believe there is value in launching this virtual clinic without delay. This will also allow further improvements to the design of the WATChmAN platform as it is being built. Therefore, this study will be divided into two stages:

Stage I: During this stage, a clinical research coordinator alongside a nurse from the Genitourinary Clinic at the Princess Margaret Cancer Centre will manually perform all the anticipated functions of the WATChmAN platform. The clinical research coordinator will be responsible for all the administrative roles of WATChmAN including sending appointment reminders and scheduling follow-up virtual appointments. The nurse will be responsible for all the clinical functionalities of the WATChmAN platform. They will manually track patients' blood and imaging test results and work closely with the Multidisciplinary Testicular Cancer Clinic physicians to ensure that all patient surveillance results are reviewed. Patients randomized to the in-person AS group will receive the traditional standard of care which includes returning to clinic to meet with physicians face-to-face to receive imaging and blood testing results.

Stage II: During stage 2 of this investigation, the WATChmAN platform will be responsible for automatically populating the virtual clinic with blood and imaging results, sending appointment reminders and scheduling follow up appointments. The responsibilities of patients randomized to the WATChmAN group will be to acknowledge these email/text appointment reminders (i.e. yes/no to being aware of upcoming appointments), checking their results virtually and scheduling follow-up appointments through the WATChmAN platform. The research coordinator and nurse will continue to oversee the WATChmAN function but will not be manually collating surveillance results (markers/imaging etc.). Patients randomized to the in-person AS group receive the traditional standard of care, returning to the clinic to meet with a physician face-to-face to receive their surveillance imaging and blood marker results.

ELIGIBILITY:
Inclusion Criteria:

* Men who are at least 18 years of age
* Can read, write, and speak English
* Have access to an electronic platform (i.e. computer, smart phone, tablet, etc.)
* Have had histologically confirmed stage 1 testicular cancer (seminoma or non- seminoma),
* Have undergone a radical orchiectomy in the last 9 months and will be/are on active surveillance under the supervision of the multidisciplinary testicular cancer clinic at Princess Margaret.
* Must be prepared to comply with the close follow-up protocol and provide informed consent

Exclusion Criteria:

* Men who have experienced metastatic disease or TCa relapse within their first 9 months of AS
* Men with inadequate computer literacy or compliance as deemed by the study team

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Efficacy | December 2017 - December 2026
  Assess the safety and efficacy of administering active surveillance for testicular cancer on a virtual platform. Specifically, patient compliance, relapse incidence, extent of relapse, burden of treatment for relapse, modes of therapy required for relapse, and distal cancer outcomes.

SECONDARY OUTCOMES:
Patient Satisfaction | December 2017 - December 2026
  Assess patient satisfaction with receiving their care virtually and with the system that administers the care.
Physician Satisfaction | December 2017 - December 2026
  Assess physician satisfaction with delivering care virtually and with the system that administers the care.
Clinic Flow Metrics | December 2017 - December 2026
  Assess how implementation of the WATChmAN virtual clinic has impacted the number of new patients seen in clinic, the CCO Wait 1 times (time from receipt of referral to first consult), physician estimations of time spent on follow-up, and examination of lost-to-follow-up rates.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Hamilton, MD, Principal Investigator — The Princess Margaret Cancer Foundation
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No